CLINICAL TRIAL: NCT04882644
Title: Effects of Aerobic Exercise on Lean Non-alcoholic Fatty Liver Disease
Brief Title: Effects of Aerobic Exercise on Lean Non-alcoholic Fatty Liver Disease (NAFLD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Qun Zhang, Professor, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NMU20212022
Record Dates: First submitted 2021-04-28; First posted 2021-05-12 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Non-alcoholic Fatty Liver Disease
Keywords: Lean NAFLD
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aerobic Exercise Intervention Group (Experimental): The subjects receive an intensive aerobic exercise for 3 months and a health education content for 12 months.
  Interventions: Behavioral: Aerobic Exercise
- Control Group (No Intervention): The subjects do not change their physical activity routine and receive a health education content for 12 months.

INTERVENTIONS:
Behavioral: Aerobic Exercise — The subjects conduct an aerobic exercise at 65-80% maximum oxygen consumption three times per week for 60 min/session (including 5 min warm-up and 5 min cool down) with treadmills, ellipticals, and rowing machine. The subjects attend health education sessions (eg, general health knowledge of NAFLD and metabolic diseases, and elements of a healthy lifestyle) monthly in the 12 months.
  Arms: Aerobic Exercise Intervention Group

SUMMARY:
NAFLD is increasingly being identified in lean individuals, especially in Chinese population. Among the NAFLD patients, the lean NAFLD accounts for 15.9%-23.0%. Previous studies showed that the lean NAFLD individuals might have a higher risk of severe hepatic disease than those obese individuals. However, the effects of aerobic exercise on the reduction of liver fat content and metabolic risk factors in lean NAFLD individuals remain unknown. In this randomized controlled trial, we will examine the effect of a 3-month exercise training (aerobic exercise) on liver fat content and metabolic risk factors in lean NAFLD individuals.

DETAILED DESCRIPTION:
The whole study is divided into four phases: recruitment phase, training phase (1 month, aim to gradually adapt patients to the target exercise intensity), implementation phase (3 months), and follow-up phase (9 months). And the subjects are randomly assigned to two groups: aerobic exercise intervention group and control group.

ELIGIBILITY:
Inclusion Criteria:

* 1. Subjects with NAFLD determined by MRI-PDFF (liver fat>5%).

  2. Subjects with BMI<23 kg/m2.

  3. Subjects with inactive exercise before.

  4. Subjects with basic abilities of understanding, communication and writing.

Exclusion Criteria:

* 1. Regular drinkers (consumed more than an average of 140 grams of ethanol per week in men and 70 grams in women during the past twelve months).

  2. Complicated with other liver diseases (i.e. acute or chronic viral hepatitis, liver cancer, liver cirrhosis, drug-induced liver diseases, and autoimmune hepatitis).

  3. Subjects with abnormal liver function (i.e. more than 3 times the upper limit of normal alanine aminotransferase and aspartate aminotransferase).

  4. Complicated with severe cardiovascular disease [i.e. myocardial infarction, arrhythmia, heart failure (New York Heart Association III or IV), uncontrolled hypertension (i.e. systolic blood pressure >180 mmHg, and/or diastolic blood pressure >100 mmHg)].

  5. Complicated with severe kidney disease or severe renal insufficiency or tumour.

  6. Currently pregnant or planning to be pregnant or breast feeding women.

  7. Participating in weight loss programs/exercise programs currently or during the past three months.

  8. Having any medical condition that would affect metabolism or limit exercise (i.e. diabetes, known hyperthyroidism or hypothyroidism).

  9. Having a medical condition that would limit exercise participation or alter heart rate during exercise or taking medication that would affect metabolism or weight loss (i.e. glucocorticoids, antithyroid drugs, hypoglycemic drugs, antihypertensive drugs).

  10. Having been doing regular physical exercise for the past three months (i.e. 3 times/week, >30 min/time).

  11. Subjects with poor adherence.

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2021-05-14 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in the liver fat content at 3 months after intervention. | 3 months
  The magnetic resonance imaging-derived proton density fat fraction (MRI-PDFF) is used to detect the liver content. An diagnosis of NAFLD is the liver fat content > 5%.
  Changes = (liver fat content at 3 months after intervention - liver fat content at baseline)

SECONDARY OUTCOMES:
Changes from baseline in body mass index (BMI) at 3/12 months after intervention. | 3 months, 12 months
  The BMI expressed in units of kg/m2 is calculated as the body weight （kilograms） divided by the square of the body height (meters) while height and weight are measured by calibrated instruments with standard protocols.
  Changes = (BMI at 3/12 months after intervention - BMI at baseline).
Changes from baseline in waist hip ratio(WHR) at 3/12 months after intervention. | 3 months, 12 months
  The WHR is calculated as the waist circumference（centimeters）divided by the hip circumference (centimeters) while waist circumference and hip circumference are measured by calibrated instruments with standard protocols.
  Changes = (WHR at 3/12 months after intervention - WHR at baseline).
Changes from baseline in abdominal fat at 3/12 months after intervention. | 3 months, 12 months
  Abdominal fat expressed in units of cm2 is detected by MRI-PDFF.
  Changes = (the values of abdominal fat at 3/12 months after intervention - the values of abdominal fat at baseline).
Changes from baseline in blood pressure at 3/12 months after intervention. | 3 months, 12 months
  Blood pressure is measured by electronic automated sphygmomanometer.
  An normal blood pressure is defined as a systolic blood pressure between 90 and 139 mmHg and a diastolic blood pressure between 60 and 89 mmHg.
  Changes = (blood pressure at 3/12 months after intervention - blood pressure at baseline)
Changes from baseline in triglycerides at 3/12 months after intervention. | 3 months, 12 months
  Triglycerides is detected by fasting blood test.
  Normal triglycerides level is less than 2.26 mmol/L.
  Changes = (triglycerides at 3/12 months after intervention - triglycerides at baseline)
Changes from baseline in total cholesterol at 3/12 months after intervention. | 3 months, 12 months
  Total cholesterol is detected by fasting blood test.
  Normal total cholesterol level is less than 5.20 mmol/L.
  Changes = (total cholesterol at 3/12 months after intervention - total cholesterol at baseline)
Changes from baseline in fasting blood glucose at 3/12 months after intervention. | 3 months, 12 months
  Fasting blood glucose is detected by fasting blood test.
  Normal fasting blood glucose level is a range of 3.90-6.10 mmol/L.
  Changes = (fasting blood glucose at 3/12 months after intervention - fasting blood glucose at baseline)
Changes from baseline in fasting insulin at 3/12 months after intervention. | 3 months, 12 months
  Fasting insulin is detected by fasting blood test.
  Normal fasting insulin level is a range of 1.8-11.8 μU/mL.
  Changes = (fasting insulin at 3/12 months after intervention - fasting insulin at baseline)
Changes from baseline in glucose level for oral glucose tolerance test (OGTT) at 3/12 months after intervention. | 3 months, 12 months
  Participants will fast for at least 10 hours before the test. After a fasting blood sample is drawn, participants will drink 75g glucose in 300 ml water within 3-5 minutes. Blood samples will be drawn at 30 min, 60min and 120 min after glucose loading to measure glucose.
  Normal glucose level for OGTT at 2 hours is <7.8 mmol/L.
  Changes = (glucose level for OGTT at 2 hours at 3/12 months after intervention - glucose level for OGTT at 2 hours at baseline)
Changes from baseline in homeostasis model assessment of insulin resistance (HOMA-IR) at 3/12 months after intervention. | 3 months, 12 months
  HOMA-IR is calculated as [fasting glucose (mmol/L)* fasting insulin (μU/mL) ] / 22.5.
  HOMA-IR < 1 signals optimal insulin sensitivity and HOMA-IR < 2.5 signals normal insulin sensitivity.
  Changes = (HOMA-IR at 3/12 months after intervention - HOMA-IR at baseline)
Changes from baseline in homeostasis model assessment of β-cell function (HOMA-β) at 3/12 months after intervention. | 3 months, 12 months
  HOMA-β is calculated as 20 x fasting insulin(μU/ml)/[fasting glucose (mmol/L) - 3.5].
  Changes = (HOMA-β at 3/12 months after intervention - HOMA-β at baseline)
Changes from baseline in the liver fat content at 12 months after intervention. | 12 months
  The magnetic resonance imaging-derived proton density fat fraction (MRI-PDFF) is used to detect the liver content. An diagnosis of NAFLD is the liver fat content > 5%.
  Changes = (liver fat content at 12 months after intervention - liver fat content at baseline)

CONTACTS AND LOCATIONS:
Overall Officials: Qun Zhang, Professor, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, China, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee S, Bacha F, Hannon T, Kuk JL, Boesch C, Arslanian S. Effects of aerobic versus resistance exercise without caloric restriction on abdominal fat, intrahepatic lipid, and insulin sensitivity in obese adolescent boys: a randomized, controlled trial. Diabetes. 2012 Nov;61(11):2787-95. doi: 10.2337/db12-0214. Epub 2012 Jun 29. PMID 22751691
- [Background] Zhang HJ, He J, Pan LL, Ma ZM, Han CK, Chen CS, Chen Z, Han HW, Chen S, Sun Q, Zhang JF, Li ZB, Yang SY, Li XJ, Li XY. Effects of Moderate and Vigorous Exercise on Nonalcoholic Fatty Liver Disease: A Randomized Clinical Trial. JAMA Intern Med. 2016 Aug 1;176(8):1074-82. doi: 10.1001/jamainternmed.2016.3202. PMID 27379904
- [Background] Houghton D, Thoma C, Hallsworth K, Cassidy S, Hardy T, Burt AD, Tiniakos D, Hollingsworth KG, Taylor R, Day CP, McPherson S, Anstee QM, Trenell MI. Exercise Reduces Liver Lipids and Visceral Adiposity in Patients With Nonalcoholic Steatohepatitis in a Randomized Controlled Trial. Clin Gastroenterol Hepatol. 2017 Jan;15(1):96-102.e3. doi: 10.1016/j.cgh.2016.07.031. Epub 2016 Aug 10. PMID 27521509
- [Background] Kistler KD, Brunt EM, Clark JM, Diehl AM, Sallis JF, Schwimmer JB; NASH CRN Research Group. Physical activity recommendations, exercise intensity, and histological severity of nonalcoholic fatty liver disease. Am J Gastroenterol. 2011 Mar;106(3):460-8; quiz 469. doi: 10.1038/ajg.2010.488. Epub 2011 Jan 4. PMID 21206486